CLINICAL TRIAL: NCT03606382
Title: Collection of Clinical Specimens From Volunteers for Assay Development
Status: Completed | Type: Observational
Sponsor: Inflammatix (Industry)
Responsible Party: Sponsor
Other Study IDs: DEV-INF-01
Record Dates: First submitted 2018-07-22; First posted 2018-07-30 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Acute Respiratory Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample collected in PAXgene tubes and Nasal Swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HostDx Fever Test — HostDx Fever test to distinguish between viral and bacterial infections
Diagnostic Test: HostDx Sepsis Test — HostDx Fever test to determine the severity of a presented, suspected infection.

SUMMARY:
This study will analyze gene expression data from various biological specimens collected from voluntary participants.

DETAILED DESCRIPTION:
Primary objective is the collection of specimens from volunteers for the development and validation of HostDx tests. The study does only encompass specimen collection - Therefore, no traditional endpoint is defined but rather the successful collection of clinical specimens is defined as the endpoint.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Able to provide informed consent

Exclusion Criteria:

* Known pregnancy
* Inability to understand instructions and comply with study related procedures

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Volunteer participants
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Collection of Specimens from Volunteers for the Development and Validation of HostDx Tests | 1 Day
  Blood collection, upper respiratory specimens including. nasal swabs, nasal washes, nasopharyngeal swabs, buccal swabs, buccal washes), sputum, saliva, urine and a skin/soft-tissue specimen (dermal).

CONTACTS AND LOCATIONS:
Locations (1):
- Inflammatix, Inc., Burlingame, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaieski DF, Mikkelsen ME, Band RA, Pines JM, Massone R, Furia FF, Shofer FS, Goyal M. Impact of time to antibiotics on survival in patients with severe sepsis or septic shock in whom early goal-directed therapy was initiated in the emergency department. Crit Care Med. 2010 Apr;38(4):1045-53. doi: 10.1097/CCM.0b013e3181cc4824. PMID 20048677
- [Background] Ferrer R, Martin-Loeches I, Phillips G, Osborn TM, Townsend S, Dellinger RP, Artigas A, Schorr C, Levy MM. Empiric antibiotic treatment reduces mortality in severe sepsis and septic shock from the first hour: results from a guideline-based performance improvement program. Crit Care Med. 2014 Aug;42(8):1749-55. doi: 10.1097/CCM.0000000000000330. PMID 24717459
- [Background] Singer M. Biomarkers in sepsis. Curr Opin Pulm Med. 2013 May;19(3):305-9. doi: 10.1097/MCP.0b013e32835f1b49. PMID 23411577
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Coburn B, Morris AM, Tomlinson G, Detsky AS. Does this adult patient with suspected bacteremia require blood cultures? JAMA. 2012 Aug 1;308(5):502-11. doi: 10.1001/jama.2012.8262. PMID 22851117
- [Background] Sweeney TE, Shidham A, Wong HR, Khatri P. A comprehensive time-course-based multicohort analysis of sepsis and sterile inflammation reveals a robust diagnostic gene set. Sci Transl Med. 2015 May 13;7(287):287ra71. doi: 10.1126/scitranslmed.aaa5993. PMID 25972003
- [Background] Sweeney TE, Wong HR, Khatri P. Robust classification of bacterial and viral infections via integrated host gene expression diagnostics. Sci Transl Med. 2016 Jul 6;8(346):346ra91. doi: 10.1126/scitranslmed.aaf7165. PMID 27384347
- [Background] Sweeney TE, Perumal TM, Henao R, Nichols M, Howrylak JA, Choi AM, Bermejo-Martin JF, Almansa R, Tamayo E, Davenport EE, Burnham KL, Hinds CJ, Knight JC, Woods CW, Kingsmore SF, Ginsburg GS, Wong HR, Parnell GP, Tang B, Moldawer LL, Moore FE, Omberg L, Khatri P, Tsalik EL, Mangravite LM, Langley RJ. A community approach to mortality prediction in sepsis via gene expression analysis. Nat Commun. 2018 Feb 15;9(1):694. doi: 10.1038/s41467-018-03078-2. PMID 29449546
- [Background] Sweeney TE, Khatri P. Benchmarking Sepsis Gene Expression Diagnostics Using Public Data. Crit Care Med. 2017 Jan;45(1):1-10. doi: 10.1097/CCM.0000000000002021. PMID 27681387